CLINICAL TRIAL: NCT04314076
Title: A Pilot Single-blind Randomized Controlled Trial to Evaluate the Safety and Feasibility of Rhythmic Auditory Stimulation for Gait Training in Persons With Multiple Sclerosis
Brief Title: Rhythmic Auditory Stimulation & Gait Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Consortium of Multiple Sclerosis Centers (Other); MedRhythms, Inc. (Industry)
Responsible Party: Principal Investigator, Francois Bethoux, MD, Chairman, Department of PM&R,, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: #19-1590
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic
Keywords: Gait analysis; Music therapy; Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: a single blind parallel-group pilot randomized controlled trial comparing rhythmic auditory stimulation (RAS) with gait training to gait training without RAS.
Who Masked: Outcomes Assessor
Masking Description: A blinded examiner will be used to perform the gait analysis, 6 minute walk , and timed 25 foot walk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait Training (GT) with Rhythmic Auditory Stimulation (RAS) (Active Comparator): Participants in this arm will complete 16 supervised gait training sessions consisting of continuous overground walking on a track for 30 minutes,with RAS
  Interventions: Other: Rhythmic auditory stimulation
- Gait training (GT) without Rhythmic Auditory Stimulation (RAS) (Other): Participants in this arm will complete 16 supervised gait training sessions consisting of continuous overground walking on a track for 30 minutes without RAS
  Interventions: Other: Gait Training

INTERVENTIONS:
Other: Rhythmic auditory stimulation — RAS, a Neurologic Music Therapy technique developed to utilize rhythm and timing cues to assist in improving the basic, intrinsic rhythmic movements of gait.
  Other Names: RAS
  Arms: Gait Training (GT) with Rhythmic Auditory Stimulation (RAS)
Other: Gait Training — Continuous overground walking on a track for 30 minutes. Gait training will primarily consist of walking exercise under the supervision of an exercise physiologist.
  Other Names: GT
  Arms: Gait training (GT) without Rhythmic Auditory Stimulation (RAS)

SUMMARY:
This study will enroll patients with Multiple Sclerosis and some difficulty with walking. The purpose of this study is to use Rhythmic Auditory Stimulation (RAS) a music therapy technique that provides rhythmic auditory cues (like a beat) to help improve a patient's movements, especially when walking.

Participants will be asked to participate in a walking program (WP) with Rhythmic Auditory Stimulation (RAS), or a WP without RAS.

DETAILED DESCRIPTION:
Rhythmic Auditory Stimulation (RAS) is a music therapy technique that provides rhythmic auditory cues (like a beat) to help improve patients' movements, especially when walking. The RAS can be delivered at a fixed tempo or interactive tempo.

The device used in this study will deliver an interactive tempo. The equipment will include a mobile device app and sensors that are attached to the participant's shoes. Headphones and smartphones will be required to use the device and will be provided to the study team and kept at the center for this study. The device is designed to use audio cues to facilitate improvements in the participant's walking speed while listening to music.

The overall purpose of this study is to assess the safety and acceptability of interactive RAS music combined with gait training in individuals with MS and walking impairment, and to gather preliminary efficacy data for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS based on 2017 revised McDonald criteria (relapsing or progressive course)
* Performs the T25FW in 8 to 30 seconds (cane(s), walking stick(s), crutch(es), or wheeled walker allowed)

Exclusion Criteria:

* Physical therapy in the past 3 months or immediate need for PT due to safety concerns (e.g. falls)
* Requires at least one seated rest during the 6 MW test
* Treatment with high-dose corticosteroids in the past 2 months or planned during the study period
* Lower extremity botulinum toxin (BT) injections for spasticity in the past 3 months, or planned during the study period
* Initiation of an oral symptomatic therapy which could affect walking in the past 4 weeks (particularly dalfampridine and medications for spasticity)
* Initiation of a new disease-modifying therapy for MS in the past 3 months
* Comorbidity compromising safe participation or affecting walking (e.g. uncontrolled cardiac or respiratory illness, musculoskeletal disorder)
* Severe hearing impairment with or without the use of hearing aids, such that the participant cannot hear the rhythmic music stimulus consistently.

Inability to walk safely to the rhythmic music stimulus during the baseline visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | through study completion, up to 16 weeks
  Adverse events will be collected throughout the study period to assess treatment safety.
Percentage of training sessions missed. | through end of treatment, up to 9 weeks
  Training session attendance will be tracked as an indicator of feasibility throughout the treatment period.

SECONDARY OUTCOMES:
Timed 25 Foot Walk | Week 0, Week 9 and week 16
  Participants are instructed to walk as fast as possible but safely on a 25-foot straight course.
6-Minute Walk | Week 0, Week 9 and week 16
  Participants are instructed to walk for 6 minutes.
Spatiotemporal gait parameters | Week 0, Week 9 and week 16
  Gait parameters at self-selected pace will be collected on an electronic walkway.
MS Walking Scale - 12 | Week 0, Week 9 and week 16
  The MSWS-12 consists of 12 items inquiring about the impact of MS on various aspects of walking. Score range is from 0 to 100, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Bethoux, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No